CLINICAL TRIAL: NCT07287020
Title: PRICE vs PEACE and LOVE in Adolescent Lateral Ankle Sprain Rehabilitation: a Prospective Comparative Study of Muscle Strength and Dynamic Balance.
Brief Title: PRICE vs PEACE and LOVE in Adolescent Lateral Ankle Sprain Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Matas Meškauskas, Pediatric Orthopedic Surgeon, Lithuanian University of Health Sciences, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MM-LSMU-LAS-Study
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Lateral Ankle Sprain; Ankle Injuries; Sprain of Lateral Ligament; Rupture of Ligaments at Ankle and Foot Level
Keywords: PRICE protocol; PEACE and LOVE protocol; Ankle sprain rehabilitation; Y-Balance Test; Biodex isokinetic testing
MeSH Terms: conditions — Ankle Injuries | interventions — Commerce

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned in a 1:1 ratio to one of two treatment groups using a computer-generated simple randomization sequence with concealed envelope allocation. Each participant received only the intervention assigned at randomization, and no crossover occurred between groups. Both groups were followed in parallel for the full study period, and outcome assessors were blinded to group assignment.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors performing ultrasound imaging, isokinetic strength testing, and Y-Balance assessments were blinded to treatment allocation. Participants and treating clinicians were not blinded due to the nature of the rehabilitation protocols.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRICE + NSAIDs (Active Comparator): Participants received the traditional PRICE protocol (Protection, Rest, Ice, Compression, Elevation) during the acute phase, including rest and limited weight-bearing for 3-5 days based on pain, cryotherapy four times daily for 15-20 minutes, compression, and limb elevation. Ibuprofen was prescribed three times daily according to body weight. No structured rehabilitation exercises were introduced during the first 1-2 weeks. Gradual return to full weight-bearing was allowed as symptoms improved, and a lace-up ankle splint was used during daily activities.
  Interventions: Behavioral: PRICE + NSAIDs protocol
- PEACE and LOVE (Active Comparator): Participants received the PEACE and LOVE rehabilitation approach (Protection, Elevation, Avoid anti-inflammatories, Compression, Education + Load, Optimism, Vascularization, Exercise). Cryotherapy and NSAIDs were avoided, with paracetamol used only for pain control. Early education on injury healing and self-management was provided. Pain-free home exercises were initiated during the first week, including elastic resistance strengthening and balance training. Progressive loading, neuromuscular exercises, aerobic conditioning, and sport-specific drills were added in subsequent phases. A lace-up ankle splint was used during daily activities.
  Interventions: Behavioral: PEACE and LOVE protocol

INTERVENTIONS:
Behavioral: PRICE + NSAIDs protocol — A conservative management approach consisting of Protection, Rest, Ice, Compression, and Elevation. Includes scheduled ibuprofen dosing according to body weight for pain and inflammation control. The intervention focuses on symptom reduction through cryotherapy, activity restriction, and edema management during the early phase of recovery.
  Arms: PRICE + NSAIDs
Behavioral: PEACE and LOVE protocol — A rehabilitation framework emphasizing Protection, Elevation, Avoidance of anti-inflammatories, Compression, and Education, followed by Load, Optimism, Vascularization, and Exercise. The intervention promotes early optimal loading, pain-free therapeutic exercise, neuromuscular training, and patient education to support tissue healing and functional recovery.
  Arms: PEACE and LOVE

SUMMARY:
This study compared two early management strategies for adolescents with first-time lateral ankle sprain: the traditional PRICE protocol (Protection, Rest, Ice, Compression, Elevation) combined with non-steroidal anti-inflammatory drugs (NSAIDs) and the PEACE and LOVE rehabilitation framework (Protection, Elevation, Avoid anti-inflammatories, Compression, Education + Load, Optimism, Vascularization, Exercise). Seventy-six participants aged 12-17 years were randomized to one of the two treatment groups and followed for 12-15 weeks. Functional recovery was assessed at three time points using isokinetic dynamometry to measure ankle inversion and eversion strength, and the Y-Balance Test to evaluate dynamic balance. The study aimed to determine whether the PEACE and LOVE approach resulted in superior improvements in neuromuscular function compared to PRICE + NSAIDs. Outcomes were analyzed as side-to-side deficits between the injured and uninjured limbs.

DETAILED DESCRIPTION:
This prospective randomized study evaluated two early management approaches for adolescents with first-time lateral ankle sprain. Participants aged 12 to 17 years who presented within 1 to 4 days of injury were randomized to either the PRICE protocol (Protection, Rest, Ice, Compression, Elevation) combined with non-steroidal anti-inflammatory drugs (NSAIDs) or the PEACE and LOVE rehabilitation framework (Protection, Elevation, Avoid anti-inflammatories, Compression, Education + Load, Optimism, Vascularization, Exercise). Randomization was performed using a computer-generated sequence with concealed envelope allocation. Outcome assessors were blinded to group assignment.

Both groups received initial protection using a lace-up ankle splint, and some participants received temporary plaster cast immobilization in the emergency department based on clinical symptoms. In the PRICE + NSAIDs group, early management focused on rest, cryotherapy, compression, elevation, and scheduled ibuprofen dosing according to body weight. Structured rehabilitation exercises were not introduced during the first 1 to 2 weeks. In the PEACE and LOVE group, cryotherapy and NSAIDs were avoided, and participants received education on tissue healing and early optimal loading. Home exercises included pain-free elastic resistance strengthening and basic balance training starting in the first week, with progressive neuromuscular and aerobic exercise in later phases.

Functional recovery was assessed at 1-2 weeks, 5-7 weeks, and 12-15 weeks after injury. Objective biomechanical outcomes included isokinetic ankle inversion and eversion strength and range of motion measured using a Biodex dynamometer at angular velocities of 60°/s and 120°/s. Dynamic balance was evaluated using the Y-Balance Test. All outcomes were analyzed as side-to-side deficits between the injured and uninjured limbs.

The primary aim of the study was to compare functional recovery between the two treatment protocols over a 12-15-week period. Secondary aims included evaluating changes in dynamic balance, assessing the influence of early immobilization on outcomes, and documenting the time course of strength and mobility restoration. The study was conducted at the Lithuanian University of Health Sciences and received ethics approval prior to initiation.

ELIGIBILITY:
Inclusion Criteria:

Age 12 to 17 years

First-time lateral ankle sprain

Presentation within 1 to 4 days after injury

No chronic ankle pain prior to the injury

No fracture except minor avulsion fractures confirmed by imaging

Ability to participate in follow-up assessments

Exclusion Criteria:

Previous ankle surgery

History of chronic ankle pain or ankle instability

Systemic diseases (e.g., inflammatory, metabolic, or autoimmune conditions)

Neurological disorders affecting lower-extremity function

Inability to perform isokinetic or balance testing

Declined informed consent by the participant or legal guardian

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2025-01-14 (Actual); Study Completion 2025-01-14 (Actual)

PRIMARY OUTCOMES:
Change in ankle inversion peak torque/body weight (%) deficit between injured and uninjured limbs at 60°/s | 1-2 weeks, 5-7 weeks, and 12-15 weeks after injury
  Ankle inversion peak torque normalized to body weight (Peak TQ/BW, %) is measured using a Biodex isokinetic dynamometer at an angular velocity of 60 degrees per second. For each assessment, peak torque values are collected for the uninjured and injured limbs and used to calculate a side-to-side deficit expressed as a percentage (uninjured minus injured limb).

SECONDARY OUTCOMES:
Change in Y-Balance Test composite score deficit between injured and uninjured limbs | 1-2 weeks, 5-7 weeks, and 12-15 weeks after injury
  Dynamic balance is assessed using the Y-Balance Test (YBT). For each limb, participants perform three maximal reach attempts in the anterior, posteromedial, and posterolateral directions, and a composite score is calculated by normalizing reach distances to limb length and multiplying by 100 percent. For each time point, a side-to-side deficit is calculated as the difference between the uninjured and injured limbs (uninjured minus injured limb). The secondary outcome is the change in this composite score deficit over time, comparing recovery between the PRICE + NSAIDs group and the PEACE and LOVE group.
Change in ankle inversion-eversion range of motion (ROM) deficit between injured and uninjured limbs | 1-2 weeks, 5-7 weeks, and 12-15 weeks after injury
  Ankle inversion and eversion range of motion (ROM, degrees) is measured using a Biodex isokinetic dynamometer at angular velocities of 60 degrees per second and 120 degrees per second. At each testing session, ROM is recorded for the uninjured and injured limbs, and a side-to-side deficit is calculated as the difference between limbs (uninjured minus injured limb). The secondary outcome is the change in ROM deficit over time at both testing velocities, comparing recovery between the PRICE + NSAIDs group and the PEACE and LOVE group.

OTHER OUTCOMES:
Change in ankle inversion peak torque/body weight (%) deficit at 120°/s | 1-2 weeks, 5-7 weeks, and 12-15 weeks after injury
  Inversion peak torque normalized to body weight (Peak TQ/BW, %) is measured using a Biodex isokinetic dynamometer at an angular velocity of 120 degrees per second. For each testing session, peak torque values are recorded for the uninjured and injured limbs, and a side-to-side deficit is calculated (uninjured minus injured limb). This outcome evaluates changes in inversion strength deficit at the higher testing velocity over time.
Change in ankle eversion peak torque/body weight (%) deficit at 60°/s and 120°/s | 1-2 weeks, 5-7 weeks, and 12-15 weeks after injury
  Ankle eversion peak torque normalized to body weight (Peak TQ/BW, %) is measured using a Biodex isokinetic dynamometer at angular velocities of 60 degrees per second and 120 degrees per second. For each velocity and at each time point, peak torque values for the uninjured and injured limbs are compared to calculate a side-to-side deficit (uninjured minus injured limb). This outcome evaluates changes in eversion strength deficit at both testing velocities over the course of rehabilitation.

CONTACTS AND LOCATIONS:
Overall Officials: Matas Meskauskas, Principal Investigator — Lithuanian University of Health Sciences; Emilis Cekanauskas, Professor, Study Director — Lithuanian University of Health Sciences
Locations (1):
- Lithuanian University of Health Sciences, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared publicly. De-identified datasets may be made available upon reasonable request to the corresponding author, subject to institutional approval and data protection regulations.

REFERENCES:
- [Background] Meškauskas M, Rutkauskas S, Misiūnienė M, Žumbakys J, Tomkevičiūtė J, Malcius D, Čekanauskas E. PRICE vs PEACE and LOVE in adolescent lateral ankle sprain rehabilitation: a prospective comparative study of muscle strength and dynamic balance.